CLINICAL TRIAL: NCT05975255
Title: Effective Dose of Remimazolam for Loss of Consciousness in Children: A Prospective Dose Finding Study
Brief Title: Dose Finding Study for Remimazolam in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2306-198-1445
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Drug Effect
Keywords: Remimazolam; Children; Dose

STUDY DESIGN:
Intervention Model Description: Sequential allocation to drug dosage according to result of previous participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): Remimazolam administration and evaluation of sedative effect
  Interventions: Drug: Remimazolam besylate

INTERVENTIONS:
Drug: Remimazolam besylate — Intravenous administration of predetermined dose of Byfavo for 30 seconds
  Other Names: Byfavo

SUMMARY:
This study aims to find effective dose of remimazolam for inducing loss of consciousness in children aged 2 to 8 years old. We will explore ED90 of remimazolam for loss of consciousness in 2 minutes after intravenous injection, via a up-and-down method with biased-coin design.

DETAILED DESCRIPTION:
We will administer remimazolam intravenously to the study participants. Remimazolam will be infused in 30 seconds to the participants, and we will wait for 2 minutes for the participants be sedated.

When a participant was not sedated in 2 minutes, dose of remimazolam in the next participant will be escalated by 0.05mg/kg. When a participant was sedated in 2 minutes, dose of remimazolam in the next participant will be decreased by 0.05mg/kg or maintained as same. The probability of decrement and maintenance will be 90% and 10% respectively. The dose of remimazolam in the first participant of the study will be 0.05mg/kg.

We will collect the results and obtain ED90 of remimazolam for loss of consciousness in children aged 2 to 8 years old.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled to undergo general anesthesia or sedation
* American Society of Anesthesiologist Physical Status of 1 or 2

Exclusion Criteria:

* Presence of Upper respiratory tract infection or any pulmonary disease
* Presence of subglottic stenosis, laryngomalacia, or tracheomalacia
* History of hypersensitivity to benzodiazepines or propofol
* History of hypersensitivity to beans or peanut
* History of seizure
* Presence of arrhythmia, tachycardia, or bradycardia
* Presence of acute closed-angle glaucoma
* Patients with unstable vital sign
* Presence of sleep apnea
* Presence of galactose intolerance, Lapp lactase deficiency, or glucose-galactose absorption disorder
* History of hypersensitivity to dextran 40
* Refusal to enroll by one or more parents or legal guardian
* Other conditions the researchers regarded as inappropriate to enroll

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Loss of consciousness | From start of remimazolam administration to 2 minute after end of administration
  Score 3 or more in the University of Michigan Sedation Scale in less than 2 minutes after administration of remimazolam besylate

SECONDARY OUTCOMES:
UMSS (University of Michigan Sedation Scale) | From start of remimazolam administration to 2 minute after end of administration
  Serial measurement of University of Michigan Sedation Scale
Heart rate | From start of remimazolam administration to 2 minute after end of administration
  Serial measurement of heart rate
Pulse oximetry | From start of remimazolam administration to 2 minute after end of administration
  Serial measurement of pulse oximetry
Noninvasive mean blood pressure | From start of remimazolam administration to 2 minute after end of administration
  Serial measurement of noninvasive mean blood pressure
Anesthetic depth | From start of remimazolam administration to 2 minute after end of administration
  Serial measurement of electroencephalogram-based anesthetic depth monitoring
Apnea | From start of remimazolam administration to 2 minute after end of administration
  Incidence of apnea after administration of remimazolam besylate

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kilpatrick GJ, McIntyre MS, Cox RF, Stafford JA, Pacofsky GJ, Lovell GG, Wiard RP, Feldman PL, Collins H, Waszczak BL, Tilbrook GS. CNS 7056: a novel ultra-short-acting Benzodiazepine. Anesthesiology. 2007 Jul;107(1):60-6. doi: 10.1097/01.anes.0000267503.85085.c0. PMID 17585216
- [Background] Gorges M, Zhou G, Brant R, Ansermino JM. Sequential allocation trial design in anesthesia: an introduction to methods, modeling, and clinical applications. Paediatr Anaesth. 2017 Mar;27(3):240-247. doi: 10.1111/pan.13088. Epub 2017 Feb 17. PMID 28211193
- [Background] Antonik LJ, Goldwater DR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part I. Safety, efficacy, and basic pharmacokinetics. Anesth Analg. 2012 Aug;115(2):274-83. doi: 10.1213/ANE.0b013e31823f0c28. Epub 2011 Dec 20. PMID 22190555